CLINICAL TRIAL: NCT06788210
Title: The Role of the Geriatric Team in Facilitating the Emergency Department (ED) Workflow for Elderly Patients: Effects on Rate of Hospitalization and on Community Health Management: A Multicentric Randomized Controlled Intervention Study
Brief Title: Geriatric Team in ED: Effects on Rate of Hospitalization and on Community Health Management of Elderly (GerED-21)
Acronym: GerED-21
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: GerED-21; 3665 (Other Grant/Funding Number: SIRER)
Record Dates: First submitted 2024-11-06; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-11

CONDITIONS: Comparative Effectiveness Research
Keywords: Elderly patients >= 75 years; Geriatric Team; CGA; Emergency room
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Intervention Model Description: The study is a multicentric interventional randomized controlled trial that involves cluster randomization, in which calendar weeks will be selected for treatment instead of patients.In the week selected as 'treatment,' the multidisciplinary team will be present in the ED and will recruit all patients who access, meet the inclusion and exclusion criteria, and provide consent to participate in the study until the required weekly number is reached. In the week selected as 'control,' patients who access and meet the inclusion and exclusion criteria will be asked for consent to participate in the study and will follow the usual care. The opulation of the study includes patients aged 75 years and older, with a Triage Risk Stratification Tool (TRST) ≥ 2, who provide consent to participate. Are excluded patients with acute pathology requiring immediate intervention in intensive areas (politrauma, urgent surgery) or who need specific pathways (Miocardial Infarction , stroke, hip fracture).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): During the weeks selected as 'control', patients who access and meet the inclusion and exclusion criteria will be asked for consent to participate in the study and will follow the usual care. An independent researcher will perform a Multidimensional assessment.
- The Geriatric Emergency Team (GET) applied CGA to identify adult patients to safely discharge (Experimental): The Geriatric Emergency Team (GET), including a geriatrician, a nurse expert in transitional care, and a social worker, conducts a front-door Comprehensive Geriatric Assessment (CGA) to identify patients who require inpatient care and those who can safely be discharged. The multidimensional assessment includes the following instruments of evaluation: SPMSQ, ADL, IADL, Charlson Comorbidity Index, Rockwood Frailty Index, GCS-5 item, number of medications, and screening for delirium (4AT). The intervention consists of counseling and information, drug therapy optimization/deprescribing, planning referral to the Center for Diagnosis of Cognitive Disorders and Dementia, contact with the patient's general practitioner, physiotherapy and walking aid prescription, social worker referral, activation of home healthcare and assistance services, transfer to a community hospital/transitional care facility, and assessment for nursing home admission.
  Interventions: Other: Multiprofessional Geriatric Emergency Team applied front-door CGA to identify patients who require inpatient care and those who can safely be discharged.

INTERVENTIONS:
Other: Multiprofessional Geriatric Emergency Team applied front-door CGA to identify patients who require inpatient care and those who can safely be discharged. — In comparison to the precedent studies, this project is characterised by some innovative aspects as regards to the design of intervention:
  1. the participation of both a geriatrician and a nurse expert in transitional care, with the consultancy of a social worker when needed, in the management of the elderly patient within ED, adds to the project a greater operational capacity of the multidimensional assessment (CGA) of planning the best care setting for the patient.
  2. The proposed CGA model is complete in the analysis of the different domains (social, clinical, functional, cognitive-affective) and achievable in this particular urgent setting.
  3. The program examines, unlike other studies, much more variables that can help to define the effectiveness of the intervention.
  4. The involvement in the network program of three main hospitals of the Emilia Romagna with a pool of elderly patients afferent to ED of about 20,000 elderly/year per hospital (2019 data prior of Sars Cov2 pandemic)
  Arms: The Geriatric Emergency Team (GET) applied CGA to identify adult patients to safely discharge

SUMMARY:
The Ger-ED Intervention study focuses on early assessment and intervention in the emergency department (ED) by a specialized geriatric team, which includes a geriatrician, a nurse with expertise in geriatrics and continuity of care from hospital to community and when necessary a social worker. The intervention model is based on Comprehensive Geriatric Assessment (CGA) and aims to improve the management and care pathways for elderly patients. Through tailored responses, the team is expected to identify the appropriate setting for each patient and coordinate with community services to facilitate a safe return home when hospitalization is avoidable, and the risks outweigh the benefits.

The purpose of this study is to evaluate the impact of this dedicated ED multidisciplinary geriatric team intervention on the quality of care for elderly patients presenting at the ED, compared to usual care.

The study is a multicentric interventional randomized controlled trial involving cluster randomization, where calendar weeks are randomized rather than individual patients.

Study Design:

During the weeks designated as 'treatment', the multidisciplinary team will be present in the ED. They will recruit all eligible patients who meet the inclusion and exclusion criteria and provide consent to participate in the study, until the required weekly number is reached.

During the weeks designated as 'control', patients who meet the inclusion and exclusion criteria and provide consent will receive the usual care.

DETAILED DESCRIPTION:
The GerED-21 study aims to introduce a multidisciplinary geriatric team model across three Northern Italian hospitals to reduce unnecessary hospitalizations among elderly emergency department (ED) patients. The Geriatric Emergency Team (GET) - comprising a geriatrician, a nurse specialized in transitional care, and a social worker - will conduct a front-door comprehensive geriatric assessment (CGA) to determine which patients require inpatient care and which can be safely discharged.

The study is planned for a 24-month duration. The first six months will focus on training team members, setting up a database, and arranging logistics within the EDs. The target population includes 624 patients aged 75 and older, admitted to the EDs of three hospitals: IRCCS AOU Policlinico di Sant'Orsola Bologna, Ospedale Maggiore AUSL Bologna, and Ospedale Maggiore AOU Parma, over 52 weeks following the start of the study at each site.

At various timepoints, data will be collected from patients, including:

Demographics: Age, sex, education level, housing status (home, sheltered facility, other hospital), cohabitation status (alone, with spouse, others), and primary caregiver.

Referral Details: Whether referred by an attending physician or direct access to the emergency room.

Multidimensional Assessment Data: Short Portable Mental Status Questionnaire (SPMSQ) , Activities of Daily Living (ADL), Instrumental Activities of Daily Living (IADL), Charlson Comorbidity Index, Rockwood Frailty Index, Geriatric Depression Scale (GDS-5 item), and number of medications.

Delirium Screening: Using the 4AT tool. ED Presentation : Date and time of presentation, clinical diagnosis (reason/condition for ED visit and ICD-9 code at discharge), triage color code (1 red, 2 orange, 3 blue, 4 green, 5 white), 3 months following ED access (including intercurrent hospitalizations).

Patients' Follow-up: Follow-up will be conducted through phone calls and record linkage with administrative data at two timepoints: A- At 7 days post-ED discharge, data on new ED visits, hospital admissions, and corresponding diagnoses according to Canadian Emergency Department Information System (CEDIS) and discharge codes (ICD-9) will be collected. B- At 30 days and 3 months post-discharge of the index ED visit for all patients, data on new ED visits, hospitalizations, functional status (Activities of Daily Living (ADL) and Instrumental Activities of Daily Living (IADL), institutionalization, and mortality will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 75 years
* Triage Risk Screening Tool (TRST) score ≥ 2
* Presence of signed informed consent

Exclusion Criteria:

* Patients with acute pathology requiring immediate intervention (polytrauma, urgent surgery)
* Patients who need specific pathway (STEMI, Stroke, Hip Fracture, patients with highly contagious diseases, for example Sars Cov2)

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 624 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-08-08 (Actual)

PRIMARY OUTCOMES:
Change the ED hospitalization rate in the intervention arm compared with the control arm | Discharge from ED at baseline access
  Expected result: >= 6% difference in hospitalization rate in patients receiving multidisciplinary evaluation compared to those following the standard care pathway.
  Measue: Proportion of patients assigned by ED to Emergency Medicine or medical/surgical ward vs. those discharged to home, facility or nursing home.

SECONDARY OUTCOMES:
Change in rate of new accesses in the ED and hospital admission | Patients participating in the study will also be asked for consent to be contacted by telephone at 7 days, 30 days and three months from access to the PS to carry out the follow-up with respect to secondary outcomes
  Change in re-attendance rate at the ED within 7 and 30 days after the index access in elderly patients discharged Measure: Proportion of patients who needed a new ED visit for the same reason/condition
Change in rate of mortality | Patients participating in the study will also be asked for consent to be contacted by telephone at 7 days, 30 days and three months from access to the PS to carry out the follow-up with respect to secondary outcomes
  Mortality rates at 30 and 90 days after index access to the ED in all patients.
  Measure:% of deaths at 30 and at 90 days in all patients after index access to the ED
Change in rate of loss of autonomy | Patients participating in the study will also be asked for consent to be contacted by telephone at 7 days, 30 days and three months from access to the PS to carry out the follow-up with respect to secondary outcomes
  Change in Activitiesof Daily Living (ADLs) score at 30 and 90 days after index access to the ED in all patients.
  Measure: ADLs score (0-6) , where the higher score means better autonomy. Change in Instrumentale Activities of Daily Living (IADLs) score at 30 and 90 days after index access to the ED in all patients.
  Measure :IADLs score (0-5) in males and (0-8) in females at 30 and 90 days after index access to the ED in all patients, where the higher score means better autonomy

CONTACTS AND LOCATIONS:
Overall Officials: Maria L Lunardelli, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No